CLINICAL TRIAL: NCT03041324
Title: A Phase I / 2, Multicenter, Open-label, Single-dose, Dose-ranging Study to Assess the Safety and Tolerability of SB-913, a rAAV2/6-based Gene Transfer in Subjects With Mucopolysaccharidosis II (MPS II)
Brief Title: Ascending Dose Study of Genome Editing by the Zinc Finger Nuclease (ZFN) Therapeutic SB-913 in Subjects With MPS II
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: All nine subjects dosed in the study have rolled over to the Long-Term Follow-up Study IVPRP-LT01 [NCT04628871]
Sponsor: Sangamo Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SB-913-1602
Record Dates: First submitted 2017-01-13; First posted 2017-02-02 (Estimated); Results first posted 2022-09-27 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Mucopolysaccharidosis II; MPS II
Keywords: MPS ll; Mucopolysaccharidosis II; Hunter syndrome; Gene Editing; Gene therapy; Zinc Finger; ZFN; SB-913; Rare; Genetic; DNA; Sangamo; Genome editing; Champions; Hunter; Gene Specific Targeted Insertion
MeSH Terms: conditions — Mucopolysaccharidosis II; Sudden Infant Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 SB-913 Starting Dose 5.00E+12 vg/kg (Experimental): A single dose of each of the three components of SB-913 [zinc finger nucleases (ZFN1, ZFN2, and hIDUA Donor)] administered via intravenous (IV) infusion.
  Interventions: Biological: SB-913
- Cohort 2 SB-913 at Next Ascending Dose 1.00E+13 vg/kg (Experimental): A single dose of each of the three components of SB-913 [zinc finger nucleases (ZFN1, ZFN2, and hIDUA Donor)] administered via intravenous (IV) infusion.
  Interventions: Biological: SB-913
- Cohort 3 SB-913 at Next Ascending Dose 5.00E+13 vg/kg (Experimental): A single dose of each of the three components of SB-913 [zinc finger nucleases (ZFN1, ZFN2, and hIDUA Donor)] administered via intravenous (IV) infusion.
  Interventions: Biological: SB-913

INTERVENTIONS:
Biological: SB-913 — Single dose of each of the 3 components of SB-913: ZFN1, ZFN2 and hIDS Donor

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability and effect on leukocyte and plasma Iduronate 2-Sulfatase (IDS) enzyme activity of ascending doses of SB-913. SB-913 is an intravenously delivered Zinc Finger Nuclease (ZFN) Therapeutic for genome editing. It inserts a correct copy of the IDS gene into the Albumin locus in hepatocytes with the goal of lifelong therapeutic production of the IDS enzyme.

DETAILED DESCRIPTION:
The objectives of the study are to provide long term expression of IDS and improve the current clinical outcome of enzyme replacement therapy (ERT) in subjects with MPS II, a recessive lysosomal storage disorder that results from mutations in the gene encoding IDS. SB-913 is a therapeutic for ZFN-mediated genome editing which will be delivered by adeno-associated virus (AAV)-derived vectors. SB-913 is intended to function by placement of the corrective copy of IDS transgene into the genome of the subject's own hepatocytes, under the control of the highly expressed endogenous albumin locus, and is expected to provide permanent, liver-specific expression of Iduronate 2-Sulfatase for the lifetime of an MPS II patient.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 5 years to 65 years of age.
* Clinical diagnosis of MPS II (based on evidence of hepatosplenomegaly, dysostosis multiplex by X-ray, valvular heart disease, or obstructive airway disease) IDS deficiency confirmed by gene sequencing.

Exclusion Criteria:

* Known to be unresponsive to ERT
* Neutralizing antibodies to AAV 2/6
* Serious intercurrent illness or clinically significant organic disease (unless secondary to MPS II)
* Receiving antiviral therapy for hepatitis B or C, or with active hepatitis B or hepatitis C or HIV 1/2
* Lack of tolerance to idursulfase treatment with significant IARs or occurrence of anaphylaxis
* Markers of hepatic dysfunction
* Creatinine ≥ 1.5 mg/dL
* Contraindication to the use of corticosteroids for immunosuppression
* Current treatment with systemic (IV or oral) immunomodulatory agent or steroid use (topical treatment allowed)
* Participation in prior investigational drug or medical device study within the previous 3 months
* Prior treatment with a gene therapy product
* Elevated or abnormal circulating α-fetoprotein (AFP)
* Weight < 20 kg at Screening Visit

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2021-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sangamo Therapeutics
Locations (5):
- United States (5):
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - NYU School of Medicine, Neurogenetics Division, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Harmatz P, Prada CE, Burton BK, Lau H, Kessler CM, Cao L, Falaleeva M, Villegas AG, Zeitler J, Meyer K, Miller W, Wong Po Foo C, Vaidya S, Swenson W, Shiue LH, Rouy D, Muenzer J. First-in-human in vivo genome editing via AAV-zinc-finger nucleases for mucopolysaccharidosis I/II and hemophilia B. Mol Ther. 2022 Dec 7;30(12):3587-3600. doi: 10.1016/j.ymthe.2022.10.010. Epub 2022 Oct 25. PMID 36299240

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The original enrollment goal was 32 subjects: Subjects with MPS II disease sequentially enrolled in age cohorts:
  age >18 (adult cohorts 1 through 4), age 12-17 (pediatric cohorts 5 and 6), and age 5-11 (pediatric cohorts 7 and 8).
  Due to the lack of observed clinical benefit, Sangamo Therapeutics, Inc. decided to stop enrollment in this study at 9 subjects, all adults in 3 cohorts. We continue to monitor the subjects in a 10-year, long-term follow-up study ST-IVPRP-LT01 (NCT04628871).
Groups:
- Experimental: Cohort 1 SB-913 Starting Dose 5.00E+12 vg/kg; Experimental: Cohort 2 SB-913 at Next Ascending Dose 1.00E+13 vg/kg; Experimental: Cohort 3 SB-913 at Next Ascending Dose 5.00E+13 vg/kg: A single dose of each of the three components of SB-913 [zinc finger nucleases (ZFN1, ZFN2, and hIDUA Donor)] administered via intravenous (IV) infusion.
Period: Overall Study
Arm/Group | Experimental: Cohort 1 SB-913 Starting Dose 5.00E+12 vg/kg | Experimental: Cohort 2 SB-913 at Next Ascending Dose 1.00E+13 vg/kg | Experimental: Cohort 3 SB-913 at Next Ascending Dose 5.00E+13 vg/kg
Started | 2 | 2 | 5
Completed | 2 | 2 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: Cohort 1 SB-913 Starting Dose 5.00E+12 vg/kg | Experimental: Cohort 2 SB-913 at Next Ascending Dose 1.00E+13 vg/kg | Experimental: Cohort 3 SB-913 at Next Ascending Dose 5.00E+13 vg/kg | Total
Number analyzed (Participants) | 2 | 2 | 5 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 5 | 9
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 2 | 2 | 5 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 1 | 2 | 5 | 8
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 5 | 9
Baseline Iduronate 2 Sulfatase (IDS) Results [Mean (Standard Deviation); unit: nmol/mL/hr] | 4.93 (1.79605) | 1.21 (0.55154) | 7.054 (3.74949) | 5.2833 (3.68909)
Baseline Urine Glycosaminoglycans (GAG) Levels [Mean (Standard Deviation); unit: (g/mol creatinine)]
  Dermatan Sulfate, Urine (g/mol creatinine) | 4.255 (1.70413) | 5.165 (1.83141) | 4.094 (0.79563) | 4.3678 (1.14354)
  Heparan Sulfate, Urine (g/mol creatinine) | 4.955 (0.24749) | 9.795 (4.16486) | 5.074 (0.76843) | 6.0967 (2.62108)
  Total GAG (g/mol creatinine) | 4.785 (1.44957) | 6.88 (0.9051) | 4.816 (2.96001) | 5.2678 (2.36252)

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) [ Time Frame: Up to 36 Months After the SB-913 Infusion
Description: Number of participants with Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) in subjects who receive SB-913 as assessed by Common Terminology Criteria for Adverse Events (CTCAE)
Time Frame: Up to 36 months after the SB-913 infusion
Population: All subjects in this study who received any portion of the SB-913 infusion
Measure: Number; unit: participants
Groups:
- Experimental: Cohort 1 SB-913 Starting Dose 5.00E+12 vg/kg; Experimental: Cohort 2 SB-913 at Next Ascending Dose 1.00E+13 vg/kg; Experimental: Cohort 3 SB-913 at Next Ascending Dose 5.00E+13 vg/kg: A single dose of each of the three components of SB-913 [zinc finger nucleases (ZFN1, ZFN2, and hIDUA Donor)] administered via intravenous (IV) infusion.
  SB-913: Single dose of each of the 3 components of SB-913: ZFN1, ZFN2 and hIDS Donor
Arm/Group | Experimental: Cohort 1 SB-913 Starting Dose 5.00E+12 vg/kg | Experimental: Cohort 2 SB-913 at Next Ascending Dose 1.00E+13 vg/kg | Experimental: Cohort 3 SB-913 at Next Ascending Dose 5.00E+13 vg/kg
Number analyzed (Participants) | 2 | 2 | 5
participants | 2 | 2 | 5

2. Secondary Outcome: Effect of SB-913 on IDS Activity
Description: Change from baseline in clinical laboratory measurement of IDS activity measured in blood, at Month 33.
Time Frame: Baseline and Month 33 after the SB-913 infusion
Population: All subjects in this study who received any dose of the SB-913 infusion
Measure: Mean (Standard Deviation); unit: nmol/mL/hr
Arm/Group | Experimental: Cohort 1 SB-913 Starting Dose 5.00E+12 vg/kg | Experimental: Cohort 2 SB-913 at Next Ascending Dose 1.00E+13 vg/kg | Experimental: Cohort 3 SB-913 at Next Ascending Dose 5.00E+13 vg/kg
Number analyzed (Participants) | 2 | 0 | 0
nmol/mL/hr | -2.6600 (3.5213) |  |

3. Secondary Outcome: Effect of SB-913 on Urine Glycosaminoglycans (GAG) Levels
Description: Change from baseline in total GAG, Dermatan Sulfate GAG, and Heparan Sulfate GAG measured in urine at Month 36
Time Frame: Baseline and 36 months after the SB-913 infusion
Population: All subjects in this study who received any dose of the SB-913 infusion
Measure: Mean (Standard Deviation); unit: g/mol creatinine
Arm/Group | Experimental: Cohort 1 SB-913 Starting Dose 5.00E+12 vg/kg | Experimental: Cohort 2 SB-913 at Next Ascending Dose 1.00E+13 vg/kg | Experimental: Cohort 3 SB-913 at Next Ascending Dose 5.00E+13 vg/kg
Number analyzed (Participants) | 2 | 1 | 5
g/mol creatinine
  Total GAG | 1.035 (0.03536) | -2.6 (NA) — For total GAG, at month 36, only one patient in cohort 2 had a sample tested for total GAG, so no standard deviation was available. | 1.734 (1.58357)
  Dermatan Sulfate Urine | -0.025 (1.18087) | -3.39 (NA) — For DS GAG, at month 36, only one patient in cohort 2 had a sample tested for DS GAG, so no standard deviation was available. | 0.262 (0.6985)
  Heparan Sulfate Urine | 1.895 (2.39709) | -7.6 (NA) — For HS GAG, at month 36, only one patient in cohort 2 had a sample tested for HS GAG, so no standard deviation was available. | 2.880 (2.91261)

4. Secondary Outcome: Annualized Frequency of Idursulfase (or Equivalent ERT) Administration.
Description: Change from baseline in annualized frequency of idursulfase (or equivalent ERT)
Time Frame: Up to 36 months after the SB-913 infusion
Population: All subjects in this study who received any dose of the SB-913 infusion
Measure: Mean (Standard Deviation); unit: Number of Infusions
Arm/Group | Experimental: Cohort 1 SB-913 Starting Dose 5.00E+12 vg/kg | Experimental: Cohort 2 SB-913 at Next Ascending Dose 1.00E+13 vg/kg | Experimental: Cohort 3 SB-913 at Next Ascending Dose 5.00E+13 vg/kg
Number analyzed (Participants) | 1 | 2 | 5
Number of Infusions | -2.8 (NA) — Only one subject in this cohort had ERT withdrawal, so no standard deviation is available. | 9.9 (25.5) | -0.5 (6.13)

5. Secondary Outcome: AAV2/6 Clearance in Plasma, Saliva, Urine, Stool, and Semen
Description: Subjects with AAV2/6 clearance in plasma, saliva, urine, stool, and semen by PCR by Week 24.
  All the subjects had AAV2/6 clearance in all the samples assessed (i.e., plasma, saliva, urine, stool, and semen) by week 24.
  Subjects were only tested until Week 24 because, by that time, they all had 3 consecutive negative tests in all body fluids.
Time Frame: Up to 36 months after the SB-913 infusion
Population: All subjects in this study who received any portion of the SB-913 infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Cohort 1 SB-913 Starting Dose 5.00E+12 vg/kg | Experimental: Cohort 2 SB-913 at Next Ascending Dose 1.00E+13 vg/kg | Experimental: Cohort 3 SB-913 at Next Ascending Dose 5.00E+13 vg/kg
Number analyzed (Participants) | 2 | 2 | 5
Participants | 2 | 2 | 5

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the subject's date of screening until their end of study visit which ranged from 24 to 36 months.
Arm/Group | Experimental: Cohort 1 SB-913 Starting Dose 5.00E+12 vg/kg | Experimental: Cohort 2 SB-913 at Next Ascending Dose 1.00E+13 vg/kg | Experimental: Cohort 3 SB-913 at Next Ascending Dose 5.00E+13 vg/kg
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/2 | 1/2 | 3/5
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Cohort 1 SB-913 Starting Dose 5.00E+12 vg/kg (N=2) | Experimental: Cohort 2 SB-913 at Next Ascending Dose 1.00E+13 vg/kg (N=2) | Experimental: Cohort 3 SB-913 at Next Ascending Dose 5.00E+13 vg/kg (N=5)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Incarcerated Umbilical Hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) — fever
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — worsening
Lacunar Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Device Dislocation (Product Issues) | 0 (0) | 0 (0) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Cohort 1 SB-913 Starting Dose 5.00E+12 vg/kg (N=2) | Experimental: Cohort 2 SB-913 at Next Ascending Dose 1.00E+13 vg/kg (N=2) | Experimental: Cohort 3 SB-913 at Next Ascending Dose 5.00E+13 vg/kg (N=5)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Aortic Stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiomegaly (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Left Atrial Dilatation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Mitral Spinal Stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Palpatations (Cardiac disorders) | 0 (0) | 1 (4) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tachypnea (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ear Congestion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Vision Blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Visual Impairment (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdomen Pain, Upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal Pain, Lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (2)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Food Poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1 (4) | 0 (0) | 1 (1)
Jejunal Stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Oesophageal Stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatic Cyst (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (2)
Impaired Healing (General disorders) | 0 (0) | 0 (0) | 1 (1)
Influenza like Illness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Prosthetic Cardiac Valve Stenosis (General disorders) | 0 (0) | 0 (0) | 1 (1)
Thirst (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hepatocellular Injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2)
Mild Fibrosis in few portal tracts (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Portal Fibrosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Seasonal Allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Bacterial Test Positive (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Blood Urine Present (Investigations) | 0 (0) | 0 (0) | 1 (1)
Ear Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Skin Candida (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (8) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 1 (2)
Incision Site Pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Post Procedural Discharge (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Post Procedural Hematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — following liver biosy
Post Procedural Vomiting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Procedural Pain (Injury, poisoning and procedural complications) | 1 (2) | 2 (3) | 2 (3)
Skin Abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 1 (1) | 2 (2) — elevated liver function test
Aspartate Aminotransferase Increased (Investigations) | 1 (1) | 1 (2) | 2 (2) — elevated liver function test
Blood Phosphorus Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood Pressure Systolic Increased (Investigations) | 0 (0) | 0 (0) | 1 (4)
Blood Thyroid Stimulating Hormone Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
CSF Glucose Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Crystals Urine Present (Investigations) | 0 (0) | 0 (0) | 2 (2)
Decreased Phosphorous (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lmphocyte Count Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Neutrophils Count Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Prothrombin Time Prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0)
Red Cell Distribution Width Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Urinary Glycosaminoglycans Increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
White Blood Cell Count Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) — worsening
Weight Decreased. (Investigations) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Cervical Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Mobility Decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle Spasms Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle Strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral Atrophy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — thinning and atrophy (noted on ct)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — transient slurred speech
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
White Matter Lesion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (3) | 1 (2)
Devise Dislocation (Product Issues) | 0 (0) | 0 (0) | 1 (1)
Foreign Body Aspiration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — aspiration from c-pap machine
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (2) | 1 (1)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Bacteriuria (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic Lesion (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal Cyst (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Scrotal Swelling (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) — worsening
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — bloody nose
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Tracheal Disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Application Site Rash (General disorders) | 0 (0) | 1 (1) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) — left mid scalp (superficial and nodular patterns)
Cold Sweat (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Rash on wrists, bilaterally (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin Abrasion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — arm
Skin Irritation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Loss Of Personal Independence In Daily Activities (Social circumstances) | 0 (0) | 0 (0) | 1 (1)
Aortic Dilatation (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) — lower left extremity
Flushing (Vascular disorders) | 0 (0) | 1 (2) | 2 (2) — during and post ert infusion
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Infusion Site Extravasation (General disorders) | 0 (0) | 0 (0) | 1 (1)
Swelling (General disorders) | 0 (0) | 0 (0) | 1 (1)
Lower Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Blood Lactate Dehydrogenase Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Device Loosening (Product Issues) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Incarcerated Umbilical Hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to the limited sample size of 9 subjects, the primary and secondary endpoints could not be analyzed, and this study could not report any conclusions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-12-12): https://cdn.clinicaltrials.gov/large-docs/24/NCT03041324/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-30): https://cdn.clinicaltrials.gov/large-docs/24/NCT03041324/SAP_001.pdf